CLINICAL TRIAL: NCT01731184
Title: Randomized Double-blind Placebo-controlled Trial: Administration of Morphine-Placebo vs. Morphine-Midazolam in Pre-hospital Traumatic Patients With Severe Acute Pain.
Brief Title: Morphine-Midazolam in Pre-hospital Traumatic Patients With Severe Acute Pain
Acronym: Morphine-Mida
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier de Cornouaille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Morphine Midazolam
Record Dates: First submitted 2012-11-13; First posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Acute Traumatic Pain
Keywords: acute traumatic pain, pre-hospital setting, Midazolam
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Midazolam (Experimental): Midazolam (Hypnovel) at 0.04 mg /kg with morphine titration (first bolus: 0.1 mg/kg then 3 mg every 5 minutes).
  Interventions: Drug: Midazolam
- Placebo (Placebo Comparator): Placebo at 0.04 mg /kg with morphine titration (first bolus: 0.1 mg/kg then 3 mg every 5 minutes).

INTERVENTIONS:
Drug: Midazolam — Midazolam (Hypnovel) at 0.04 mg /kg with morphine titration (first bolus: 0.1 mg/kg then 3 mg every 5 minutes).
  Other Names: Midazolam (hypnovel)
  Arms: Midazolam

SUMMARY:
Administration of midazolam with morphine in patients with severe acute pain is a routine practice in the management of pre- and post-operative patients but has not been evaluated in pre-hospital setting. The investigators aim to evaluate the co-analgesic effect of midazolam in the pre-hospital management of traumatic patients with severe acute pain.

In a multicenter prospective randomized double-blind placebo-controlled trial, the investigators would like to compare the analgesic effect and safety of the intravenous morphine 0.10 mg/kg and midazolam 0.04 mg/kg with the intravenous morphine 0.10 mg/kg and placebo in pre-hospital traumatic adults. Assessment will be done at the baseline using a validated numeric rating scale (NRS).

The primary outcome will be the proportion of patients with a pain score less than or equal to 3 after 20 minutes. The secondary outcomes will be in between-group comparison of: the treatment safety, pain score every 5 minutes during 30 minutes and the total morphine dose required until obtaining a pain score less than or equal to 3.

DETAILED DESCRIPTION:
Patient will be included in pre-hospital setting. They must have an acute pain NRS greater than or equal to 6 from a traumatic origin. The participation of the study for each patient will be the time of the pre-hospital setting. The study will stop when the patient arrives at the hospital.

Patient will be randomized after obtaining an informed consent. Then, the nurse will administered intravenous morphine 0.10 mg/kg and midazolam 0.04 mg/kg or intravenous morphine 0.10 mg/kg and placebo.

Only the nurse will be aware of the treatment received by the patient. Every 5 minutes, life constants and pain score will be recorded on the case report form.

Assessment will be done at the baseline using a validated numeric rating scale. The primary outcome will be the proportion of patients with a pain score less than or equal to 3 after 20 minutes. The secondary outcomes will be in between-group comparison of: the treatment safety, pain score every 5 minutes during 30 minutes and the total morphine dose required until obtaining a pain score less than or equal to 3.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old
* conscient with spontaneous ventilation
* acute pain with an traumatic origin : pain escape superior or egal to 6/10
* taking care by French reanimation and urgency mobile services (Smur).

Exclusion Criteria:

* younger than 18 years old or older than 70 years old
* chronical respiratory insufficiency
* severe hepatocellular insufficiency,
* myasthenia
* known allergy to morphine or benzodiazepin,
* already treated for a chronical pain,
* pregnant women
* treated by morphine
* patient unable to evaluate his/her pain
* any acute and severe hemodynamic, respiratory or neurologic deficiency
* needed an local analgesia
* patient who received an other antalgic treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-11; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Pain score | 20 minutes
  The primary outcome was the proportion of patients with a pain score less than or equal to 3 after 20 minutes

SECONDARY OUTCOMES:
pain evolution | every 5 minutes and at the end of the study
  The secondary outcomes were in between-group comparison of:
  - pain score every 5 minutes during 30 minutes
Safety | during all the study
  The secondary outcomes were in between-group comparison of:
  - The treatment safety
Morphine total dose | During all the study
  The secondary outcomes were in between-group comparison of:
  - The total morphine dose required until obtaining pain score less than or equal to 3

CONTACTS AND LOCATIONS:
Overall Officials: Yannick AUFFRET, Dr, Principal Investigator — Centre Hospitalier intercommunal de Cornouaille
Locations (4):
- France (4):
  - CHU de Brest, Brest
  - CH de Carhaix, Carhaix-Plouguer
  - CHU de Nantes, Nantes
  - Centre Hpistalier Intercommunal de Cornouaille, Quimper

REFERENCES:
- [Derived] Auffret Y, Gouillou M, Jacob GR, Robin M, Jenvrin J, Soufflet F, Alavi Z. Does midazolam enhance pain control in prehospital management of traumatic severe pain? Am J Emerg Med. 2014 Jun;32(6):655-9. doi: 10.1016/j.ajem.2014.01.048. Epub 2014 Feb 4. PMID 24613655